CLINICAL TRIAL: NCT00931671
Title: Effects of Task-Oriented Aerobic Exercise Training on Cardiorespiratory Fitness and Cerebral Blood Flow in Chronic Stroke Patients
Brief Title: Task-Oriented Aerobic Exercise Training in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, National Taiwan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200710039R
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Cerebrovascular Accident
Keywords: Physical fitness; Cerebral circulation; Walking
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other): Exercise
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — aerobic exercise training
  Other Names: Exercise

SUMMARY:
The study is designed to investigate (1) the effects of task-oriented aerobic exercise training on cardiorespiratory fitness, cerebral blood flow, oxygenation, functional performance, and physical activity in patients with chronic stroke. (2) the association between outcomes

ELIGIBILITY:
Inclusion Criteria:

* poststroke duration > 6 months
* MMSE > 22

Exclusion Criteria:

* severe cardiovascular disease
* depression
* dementia
* other disease affect the testing of the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
symptom-limited exercise test | 12 wks

SECONDARY OUTCOMES:
transcranial Doppler measurement | 12 wks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan